CLINICAL TRIAL: NCT05927740
Title: The Efficacy of Hyperemesis Gravidarum on Macular Thickness, Corneal Thickness and Intraocular Pressure in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batman Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erhan Okuyan,M.D, Obstetrics and Gynecology specialist, Batman Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020-5
Record Dates: First submitted 2023-06-17; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Corneal Dystrophy; Macular Dystrophy; Hyperemesis Gravidarum - Severe
MeSH Terms: conditions — Corneal Dystrophies, Hereditary; Macular Degeneration

STUDY DESIGN:
Intervention Model Description: 2 groups ( group 1 hyperemesis gravidarum ) (group 2 control group)
Who Masked: Participant
Masking Description: 110
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 ( Hyperemesis gravidarum ) (Other): 55 hyperemesis gravidarum patient (11-14th gestational week of pregnancy)
  Interventions: Diagnostic Test: Optic coherence tomography
- 2( Control group) (Other): 55 healthy pregnant women (11-14th gestational week of pregnancy)
  Interventions: Diagnostic Test: Optic coherence tomography

INTERVENTIONS:
Diagnostic Test: Optic coherence tomography — Every participant was subjected to a comprehensive ophthalmologic examination which included measuring auto-refraction (average of three values, Topcon Autorefractometer model KM 8900, Japan), uncorrected visual acuity with cycloplegic refraction (with 0.5% cyclopentolate HCl), and IOP in millimeters of mercury (mmHg, Goldmann applanation tonometer). Moreover, slit-lamp biomicroscopy (HaagStreit, Bern, Switzerland) was performed, concentrating on potential corneal scarring and/or lenticular opacities.

SUMMARY:
Aim

Physiological changes in intraocular pressure as well as in the cornea and macula may occur during pregnancy.

In the literature, there are limited data on ocular findings in hyperemesis gravidarum. Therefore, we have decided to investigate the effect of hyperemesis gravidarum on macular thickness, corneal thickness and intraocular pressure (IOP).

DETAILED DESCRIPTION:
A total of 110 people, 55 of whom were diagnosed with hyperemesis gravidarum and 55 of whom were in the control group, were included in the study. The inclusion criteria for the study were as follows: First trimester (8-14 weeks of gestation) pregnancy with positive fetal heartbeat and no history of systemic disease; no continuous use of medication; diagnosis of hyperemesis gravidarum (ketonuria and weight > 3 kg or 5% of the body) and the occurrence of less than three vomiting attacks per day with loss of weight; body mass index (BMI) within normal limits; being between the ages of 18 and 40; not drinking alcohol or smoking. A total of 94 patients, 40 of whom were diagnosed with hyperemesis gravidarum and 54 healthy pregnant women, were divided into two groups by recording their age, BMI, laboratory and eye findings.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the study;

  * First trimester (8-14 weeks of gestation) pregnancy with positive fetal heartbeat and no history of systemic disease ,
  * no history of continuous drug use,
  * Diagnosis of hyperemesis gravidarum (ketonuria and weight >3 kg or 5% of the body) The occurrence of >3 vomiting attacks per day with loss of weight,
  * Body mass index (BMI) within normal limits,
  * Being between the ages of 18-40 ,
  * not drinking alcohol or smoking,
  * not using any vitamins or supplements use during the study

Exclusion Criteria:

* Any patient who did not meet the inclusion criteria was excluded from the study.
* Patients who participated in the study but later gave up

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female pregnant women
Enrollment: 110 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-02-13 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Take precautions of the effect of hyperemesis gravidarum on eye health | Healthy pregnant women and pregnant women diagnosed with Hyperemesis gravidarum between 6-14 weeks; eye examination findings were immediately recorded in the system. (within 1 day)
  The first-line treatment of Hyperemesis gravidarum (HG) patients ( 6 -14 th weeks of pregnant women ) is fluid depletion and antiemetic therapy, but in severe HG, sepsis, thrombosis secondary to parenteral nutrition, and, albeit rare, Wernicke's encephalopathy (WE). This condition (WE), which is defined as a sign of optic disc swelling that causes a diagnostic dilemma in pregnancy, can be diagnosed with a high index of suspicion by clinical signs and radiological evidence, and generally, patients experience rapid improvement in clinical symptoms with intravenous thiamine therapy. For all this reason, it is extremely important to take necessary precautions for obstetricians. Our primary outcome is to compare the macular thickness and corneal thickness of HG patients participating in the study with normal healthy pregnant women using Optic coherancetomography.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Okuyan, Principal Investigator — Batman Training and Research Hospital
Locations (1):
- Batman education adn research hospital, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Available for the journal administrator